CLINICAL TRIAL: NCT05202509
Title: Placebo Controlled, Double Blind, Randomized Cardiovascular Outcome Study to Evaluate the Effect of 10 mg Obicetrapib in Participants With ASCVD Not Adequately Controlled Despite Maximally Tolerated Lipid Modifying Therapies
Brief Title: Cardiovascular Outcome Study to Evaluate the Effect of Obicetrapib in Patients With Cardiovascular Disease
Acronym: PREVAIL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-8995-304
Record Dates: First submitted 2021-11-22; First posted 2022-01-21 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Placebo-Controlled, Double-Blind, Randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching placebo to active
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- obicetrapib 10mg (Experimental): one 10mg tablet, once daily.
  Interventions: Drug: Obicetrapib
- Placebo (Placebo Comparator): one placebo tablet, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Obicetrapib — 10mg obicetrapib tablet
  Arms: obicetrapib 10mg
Drug: Placebo — Placebo tablet to resemble obicetrapib
  Arms: Placebo

SUMMARY:
This study will be a placebo-controlled, double-blind, randomized, phase 3 study in participants with Atherosclerotic Cardiovascular Disease (ASCVD) who are not adequately controlled despite maximally tolerated lipid-lowering therapy.

DETAILED DESCRIPTION:
This study will be a placebo-controlled, double-blind, randomized, phase 3 study to evaluate the effect of 10mg Obicetrapib in participants with Atherosclerotic Cardiovascular Disease (ASCVD) who are not adequately controlled despite maximally tolerated lipid-lowering therapy to reduce the risk of cardiovascular death, myocardial infarction, stroke and non-elective coronary revascularization. The PREVAIL Study

ELIGIBILITY:
Inclusion Criteria:

* Males & females ≥ 18 years age.
* Established ASCVD including:
* Coronary artery disease
* Cerebrovascular disease
* Peripheral Artery disease
* On maximally tolerated lipid-modifying therapy
* Fasting LDL-C ≥ 55 mg/dL
* Fasting triglycerides < 400 mg/dL
* Estimated glomerular filtration rate ≥ 30 mL/min

Exclusion Criteria:

* New York Heart Association class III or IV heart failure or left ventricular ejection fraction < 30%
* Have been hospitalized for Heart Failure within 5 years prior to screening
* Had non-fatal MI, non-fatal stroke, non-elective coronary revascularization and/or hospitalization for unstable angina or chest pain within past 3 months prior to screening
* Uncontrolled hypertension
* Diagnosis of homozygous familial hypercholesterolemia (HoFH)
* Active liver disease
* HbA1c ≥10%
* Thyroid Stimulating Hormone (TSH) > 1.5 times upper limit normal
* Creatine kinase > 3 times upper limit normal
* History of malignancy with surgery in past 3 years
* History of alcohol or drug abuse within past 5 years
* Received treatment with investigational product or device within past 30 days excluding Coronavirus treatment or vaccine
* Known allergy to study drug
* Participated in previous obicetrapib trial
* Taking gemfibrozil within 30 days screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9541 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Effect (MACE) | 30 months after last participant randomized
  To evaluate the effect of obicetrapib on the risk of MACE

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ditmarsch, MD, Study Director — NewAmsterdam Pharma
Locations (591):
- United States (199):
  - Advanced Cardiovascular LLC, Alexander City, Alabama
  - Ascension - Cardiology Specialists of Birmingham, Birmingham, Alabama
  - Central Alabama Research, Birmingham, Alabama
  - Cardiovascular Associates of the Southeast, LLC, Birmingham, Alabama
  - Eastern Shore Research Institute, LLC, Fairhope, Alabama
  - The Heart Center Research, Huntsville, Alabama
  - Mobile Heart Specialists, Mobile, Alabama
  - Syed Research Consultants, Muscle Shoals, Alabama
  - Syed Research Consultants, Sheffield, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Clinical Research Institute of Arizona, LLC, Sun City West, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - NEA Baptist clinic, Jonesboro, Arkansas
  - Cardiology and Medicine Clinic, Little Rock, Arkansas
  - Advanced Research Center, Anaheim, California
  - Westside Medical Associates of Los Angeles, Beverly Hills, California
  - Hope Clinical Research LLC, Canoga Park, California
  - Titan Medical Research - Oceanside, Encinitas, California
  - Clinical Trials Research, Lincoln, California
  - Torrance Clinical Research Institute Inc., Lomita, California
  - American Institute of Research, Los Angeles, California
  - Amicis Research Center-Northridge, Northridge, California
  - Amicis Research, Northridge, California
  - Valley Clinical Trials, Inc, Northridge, California
  - Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center, Torrance, California
  - Cardiology Associates of Fairfield County, Norwalk, Connecticut
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Clearwater Cardiovascular and Interventional Consultants, Clearwater, Florida
  - Innovative Research of West Florida, Clearwater, Florida
  - Avail Clinical Research, DeLand, Florida
  - Invesclinic, Fort Lauderdale, Florida
  - Qway Research, Hialeah, Florida
  - New Generation of Medical Research, Hialeah, Florida
  - East Coast Institute for Research, Jacksonville, Florida
  - East Coast Institute for Research - Jacksonville Monroe St, Jacksonville, Florida
  - East Coast Institute for Research - Jacksonville University Blvd, Jacksonville, Florida
  - East Coast Institute for Research - Perimeter Park Court, Jacksonville, Florida
  - East Coast Institute for Research- Lake City, Lake City, Florida
  - Columbus Clinical Services, Miami, Florida
  - Finlay Medical Research Corp, Miami, Florida
  - A+ Research Inc, Miami, Florida
  - Ezy Medical Research, Miami, Florida
  - ProLive Medical Research, Miami, Florida
  - Med Research of Florida, LLC, Miami, Florida
  - New Generation of Medical Research - Naples, Naples, Florida
  - Advanced Research Institute Inc, New Port Richey, Florida
  - Ocala Research Institute, Ocala, Florida
  - Ormond Beach Clinical Research LLC, Ormond Beach, Florida
  - Headlands Research, Sarasota, Florida
  - BayCare Health System, Tampa, Florida
  - JSV Clinical Research Study, Inc, Tampa, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - East Coast Institute for Research - Canton, Canton, Georgia
  - Atlanta Heart Specialists, Cumming, Georgia
  - Alta Pharmaceutical Research Center, Dunwoody, Georgia
  - Cardiology Care Clinic of Lake Oconee, Eatonton, Georgia
  - NSC Research, Johns Creek, Georgia
  - Endocrine Research Solutions, Inc, Roswell, Georgia
  - Javara Inc - SouthCoast Health, Savannah, Georgia
  - Herman Clinical Research, Suwanee, Georgia
  - Biofortis, Inc, Addison, Illinois
  - Northwest Heart Clinical research, Arlington Heights, Illinois
  - IMA Clinical Research, PC, Chicago, Illinois
  - Clinical Investigation Specialists, Gurnee, Illinois
  - Apex Medical Research, Hazel Crest, Illinois
  - Advocate Health and Hospitals Corporation, Oakbrook Terrace, Illinois
  - Community Health Network-Anderson, Anderson, Indiana
  - Midwest Cardiovascular Research and Education Foundation, Elkhart, Indiana
  - Community Health Network, Indianapolis, Indiana
  - ASHA Clinical Research - Munster, LLC, Munster, Indiana
  - Cardiovascular Research of Northwest Indiana, LLC, Munster, Indiana
  - West Broadway Clinic, Council Bluffs, Iowa
  - The Iowa Clinic - Cardiovascular Services, Des Moines, Iowa
  - Hutchinson Clinic, Hutchinson, Kansas
  - Kansas Nephrology Research Institute, Wichita, Kansas
  - West Houston Area Clinical Trial Consultants, Wichita, Kansas
  - The Research Group of Lexington, LLC, Lexington, Kentucky
  - Louisville Metabolic and Atherosclerosis Research Center (L-MARC), Louisville, Kentucky
  - Research Integrity, Owensboro, Kentucky
  - Cambridge Medical Trials, Alexandria, Louisiana
  - Cardiovascular Associates Research, LLC - Covington, LA, Covington, Louisiana
  - Louisiana Heart Center, Slidell, Louisiana
  - Clinical Trials of America, West Monroe, Louisiana
  - Southern Clinical Research, LLC, Zachary, Louisiana
  - Northeast Cardiology Associates, Bangor, Maine
  - Javara Inc - Healthy Steps, Chevy Chase, Maryland
  - Medstar Health Research Institute, Hyattsville, Maryland
  - Optimal Research, LLC, Rockville, Maryland
  - Mass General Brigham Pentucket Medical Associates - Haverhill, Haverhill, Massachusetts
  - ActivMed Practices and Research - Methuen, Methuen, Massachusetts
  - BTC of New Bedford, New Bedford, Massachusetts
  - Aa Mrc, Llc, Flint, Michigan
  - Healthy Heart Cardiology, Grand Rapids, Michigan
  - McLaren Macomb Regional Medical Center, Mount Clemens, Michigan
  - Advanced Cardiology Associates, Rochester Hills, Michigan
  - Revival Research Institute, Southgate, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - Arcturus Healthcare, Troy, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Heart and Vascular Center at Methodist Hospital, Saint Louis Park, Minnesota
  - IMA Clinical Research - St. Louis, MO, St Louis, Missouri
  - St. Louis Heart and Vascular Cardiology, St Louis, Missouri
  - Montana Medical Research, Inc., Missoula, Montana
  - Meridian Clinical Research- Lincoln, NE, Lincoln, Nebraska
  - Sierra Clinical Research, Las Vegas, Nevada
  - AB Clinical Trials, Las Vegas, Nevada
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Advanced Heart Care, LLC, Bridgewater, New Jersey
  - Inspira Medical Centers, Mullica Hill, New Jersey
  - Cardio Metabolic Institute, Somerset, New Jersey
  - New Mexico Clinical Research & Osteoporosis Center Inc., Albuquerque, New Mexico
  - Mid-Hudson Medical Research, PLLC - New Windsor, New Windsor, New York
  - IMA Clinical Research PC and Affiliates- New York, NY, New York, New York
  - DiGiovanna Institute for Medical Education and Research, North Massapequa, New York
  - Saratoga Clinical Research, Saratoga Springs, New York
  - Chear Center LLC, The Bronx, New York
  - Meridian Clinical Research- Endwell, NY, Vestal, New York
  - Southgate Medical Group, West Seneca, New York
  - Great Lakes Medical Research, LLC, Westfield, New York
  - Javara Inc - Wake Forest Health Network Family Physicians - Sunset Avenue, Asheboro, North Carolina
  - Cary Research Group, LLC, Cary, North Carolina
  - The Presbyterian Hospital DBA Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Javara Inc - Tryon Medical Partners LLC, Charlotte, North Carolina
  - Moses H. Cone Memorial Hospital Operating Corporation d/b/a Cone Health, Greensboro, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - Clinical Trials of America, LLC - Lenoir, NC, Lenoir, North Carolina
  - Diabetes and Endocrinology Consultants, P.C, Morehead City, North Carolina
  - Burke Primary Care, Morganton, North Carolina
  - Pinehurst Medical Clinic, Inc., Pinehurst, North Carolina
  - Piedmont Healthcare - Statesville, Statesville, North Carolina
  - Wilmington Health Associates, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Meridian Clinical Research - Cincinnati, OH, Cincinnati, Ohio
  - Meridian Clinical Research - Springfield, OH, Cincinnati, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - Nexgen Research, Lima, Ohio
  - SV Research, Marion, Ohio
  - Advanced Medical Research (AMR), Maumee, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Lynn Health Science Institute - East, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Abington Medical Specialists, P.C. dba AMS Cardiolog, Horsham, Pennsylvania
  - Preferred Primary Care Physicians Group - Pleasant Hills, Pittsburgh, Pennsylvania
  - Frontier Clinical Research, Smithfield, Pennsylvania
  - Penn State Health Medical Group- Berks Cardiology, Wyomissing, Pennsylvania
  - Clinical Research Collaborative, LLC, Cumberland, Rhode Island
  - Piedmont Research Partners, LLC, Fort Mill, South Carolina
  - South Carolina Clinical Research LLC, Orangeburg, South Carolina
  - Hillcrest Clinical Research, Simpsonville, South Carolina
  - Monument Health Clinical Research, a department of Monument Health Rapid City Hospital, Inc, Rapid City, South Dakota
  - Chattanooga Research & Medicine, PLLC, Chattanooga, Tennessee
  - Stern Cardiovascular Foundation, Inc, Germantown, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - Cardiovascular Research of Knoxville, Powell, Tennessee
  - PharmaTex Research, LLC, Amarillo, Texas
  - Central Texas Clinical Research, Austin, Texas
  - Accelemed Research Institute, Austin, Texas
  - Private Practice - O. Alejandro Brusco, MD FACE PA, Corpus Christi, Texas
  - Javara Inc - Bridge Creek Family Medicine, Cypress, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - Texas Health Research & Education Institute, Dallas, Texas
  - South Texas Research Institute, Edinburg, Texas
  - David Turbay, MD, PLLC, El Paso, Texas
  - Javara Inc - Texas Health Care Family Physicians, Fort Worth, Texas
  - Valley Institute of Research - Fort Worth, Fort Worth, Texas
  - Mt. Olympus Medical Research, Friendswood, Texas
  - East Texas Cardiology, PA, Houston, Texas
  - Angiocardiac Care of Texas, Houston, Texas
  - Texas Heart Institute, Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - BioStar Clinical Research, Houston, Texas
  - Texas Center for Drug Development, Houston, Texas
  - West Houston Area Clinical Trial Consultants, LLC, Katy, Texas
  - Milton Haber, M.D, Laredo, Texas
  - North Hills Medical Research, Inc., North Richland Hills, Texas
  - Tapia Internal Medicine Clinic, Paris, Texas
  - Linq Research, LLC, Pearland, Texas
  - Styde Research, Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - San Antonio Premier Internal Medicine, San Antonio, Texas
  - Bandera Family HealthCare Research, LLC (BFHC), San Antonio, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Stephenville Medical & Surgical Clinic, Stephenville, Texas
  - Javara Inc - Highland Woods Health, The Woodlands, Texas
  - Alpine Research Organization, Inc., Clinton, Utah
  - Physicians' Research Options (PRO), Draper, Utah
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Burke Internal Medicine & Research, Burke, Virginia
  - Carient Heart & Vascular, Manassas, Virginia
  - York Clinical Research LLC, Norfolk, Virginia
  - Dominion Medical Associates, Richmond, Virginia
  - MultiCare Institute for Research and Innovation- Tacoma, Tacoma, Washington
  - Universal Research Group LLC, Tacoma, Washington
  - Prevea Health, Green Bay, Wisconsin
  - Clinical Investigation Specialists, Kenosha, Wisconsin
- Australia (15):
  - Royal Adelaide Hospital, Adelaide
  - Flinders Medical Centre, Bedford Park
  - Campbelltown Hospital, Campbelltown
  - The Prince Charles Hospital, Chermside
  - Monash Health, Clayton
  - Bridge Family Practice, Halls Creek
  - Austin Health, Heidelberg
  - Baker Heart and Diabetes Institute, Melbourne
  - The Alfred Hospital, Melbourne
  - Redcliffe Hospital, Redcliffe
  - Western Health, Saint Albans
  - Griffith University, Southport
  - Wollongong Hospital (Illawarra Shoalhaven Local Health District), Wollongong
  - The Queen Elizabeth Hospital (TQEH) - SA Health, Woodville South
  - Dr Heart Pty Ltd at Cholesterol Care Australia, Woolloongabba
- Bulgaria (35):
  - MHAT Aytos EOOD Department of Internal Diseases, Aytos
  - Medical Center Doctor Staykov EOOD, Burgas
  - UMHAT Deva Maria, Burgas
  - Medical Center Viva Feniks, Dobrich
  - MHAT Sveti Ivan Rilski, Gorna Oryahovitsa
  - MHAT Haskovo AD, Haskovo
  - MHAT City Clinic - Sveti Georgi EOOD, Montana
  - Medical Center - Cordis OOD, Pleven
  - MHAT Heart and Brain Pleven, Pleven
  - Medical Center for Rehabilitation and Sports Medicine I - Plovdiv EOOD, Plovdiv
  - UMHAT Sveti Georgi EA, Plovdiv
  - Medical Center Rusemed EOOD, Rousse
  - SHATC Medica Cor EAD, Rousse
  - Multiprofile Hospital for Active Treatment (MHAT)- Silistra, Silistra
  - MHAT Dr. Ivan Seliminski AD, Sliven
  - Medical Center for Specialized Medical Help in Cardiovascular Diseases OOD, Sofia
  - MHAT Sveta Sofia EOOD, Sofia
  - Diagnostic and Consulting Center 22 - Sofia, Sofia
  - DCC "Ascendent", Sofia
  - Diagnostic consultative center 24, Sofia
  - National Multiprofile Transport Hospital Tsar Boris Treti - Cardiology Clinic, Sofia
  - Medical Centre Medcross, Sofia
  - Diagnostic Consulting Center Convex EOOD, Sofia
  - MC Doctor Kalchev OOD, Sofia
  - "Medical Center Medic" OOD, Sofia
  - Multiprofile Hospital for Active Treatment National Cardiology Hospital, Sofia
  - CardioArt Medical Center, Stara Zagora
  - Medical Center Zara - Med, Stara Zagora
  - UMHAT Prof. Dr. Stoyan Kirkovich, Stara Zagora
  - Diagnostic Consultative Center Chaika, Varna
  - Medical Center Plazmamed Clinic, Varna
  - Specialized Hospital for Active Treatment of Cardiology, Varna
  - Medical Center Medica Plus OOD, Veliko Tarnovo
  - Medical Center Nevromedics, Veliko Tarnovo
  - Medical Center Velingrad 2017 EOOD, Velingrad
- Canada (18):
  - Medical Arts Health Research Group - Kamloops, Kamloops, British Columbia
  - Medical Arts Health Research Group - North Vancouver, North Vancouver, British Columbia
  - The Medical Arts Health Research Group - Penticton, Penticton, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - LMC Diabetes & Endocrinology Ltd. - Thornhill, Concord, Ontario
  - Dr. James Cha, Oshawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - KMH Cardiology & Diagnostic Centres - Hamilton, Stoney Creek, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - CardioVasc HR, Saint-Jean-sur-Richelieu, Quebec
  - Centre intégré universitaire de santé et de services sociaux (CIUSSS) de l'Estrie -Centre hospitalier universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec
  - Diex Recherche Trois-Rivieres, Inc, Trois-Rivières, Quebec
  - Diex Recherche Victoriaville, Victoriaville, Quebec
  - Brampton Clinical Trials, Brampton
  - Centre de recherche clinique de Laval, Laval
  - KMH Cardiology & Diagnostic Centres - Mississauga, Mississauga
  - Institut Universitaire de Cardiologie et de Pneumologie De Quebec, Québec
  - Discovery Clinical Services, Ltd, Victoria
- China (20):
  - Peking University First Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - The First People's Hospital of Changde City, Changde
  - The Second People's Hospital of Changzhou, Changzhou
  - Affiliated Hospital of Chifeng University, Chifeng
  - Daqing People's Hospital, Daqing
  - Shunde Hospital of Southern Medical University, Foshan
  - Guangdong Provincial People's Hospital, Guangzhou
  - Heilongjiang Provincial Hospital, Harbin
  - The First Affiliated Hospital of Nanyang Medical College - 2nd site, Nanyang
  - The First affiliated Hospital of Nanyang Medical College, Nanyang
  - Ningbo First Hospital, Ningbo
  - Panjin Liaoyou Gem Flower Hospital, Panjin
  - Pingxiang People's Hospital, Pingxiang
  - People's Hospital of Tianjin, Tianjin
  - Tianjin Fourth Central Hospital, Tianjin
  - Xi'an Gaoxin Hospital, Xi'an
  - Xianyang Hospital of Yan 'an University, Xianyang
  - The Third Affiliatied Hospital of Xinxiang Medical University, Xinxiang
  - Zibo City Linzi District People's Hospital, Zibo
- Croatia (5):
  - General Hospital Karlovac, Karlovac
  - Special Hospital for Medical Rehabilitation Krapinske Toplice, Krapinske Toplice
  - General Hospital Dr Josip Bencevic, Slavonski Brod
  - Polyclinic Solmed, Zagreb
  - University Hospital Center Zagreb, Zagreb
- Czechia (20):
  - Hornicka nemocnice s poliklinikou Bilina s.r.o., Bílina
  - Medicus Services SRO, Brandýs nad Labem
  - Centrum pro zdravi - kardiologie s.r.o., Brno
  - Kardiologicka ambulance Brno s.r.o., Brno
  - Amkardia sro, Brno
  - Nemocnice Havlickuv Brod, p.o., Havlíčkův Brod
  - Cevni ambulance - MATMED s.r.o., Hodonín
  - MUDr. Tomas Edelsberger - diabetologicka ambulance, Krnov
  - Lunacor s.r.o. - Centrum pro choroby srdce a cev, Kroměříž
  - KARDIOLOGIE - LIBEREC s.r.o., Liberec
  - InterKardio ML s.r.o., Mariánské Lázně
  - Edumed s.r.o., Náchod
  - PreventaMed s.r.o., Olomouc
  - CCR Ostrava s.r.o., Ostrava
  - Lunacor, s.r.o. - Centrum pro choroby srdce a cev - Otrokovice, Otrokovice
  - Kardiologie COR s.r.o., Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultní nemocnice v Motole, Prague
  - Ustredni vojenska nemocnice, Prague
  - Krajska nemocnice T. Bati, Zlín
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - Bispebjerg Hospital, Copenhagen
  - Amager Hospital, Copenhagen
  - Sydvestjysk Hospital, Esbjerg
  - Godstrup Regional Hospital (Gødstrup), Herning
  - Viborg Regional Hospital, Viborg
- Finland (3):
  - StudyCor Oy, Jyväskylä
  - Satucon Oy Kuopio, Kuopio
  - Turku University Hospital, Turku
- Georgia (19):
  - Health Ltd, Batumi
  - JSC Evex Hospitals - Batumi Referral Hospital, Batumi
  - Kutaisi Primary Health Care Center #1, Kutaisi
  - Bokhua Memorial Cardiovascular Center LTD, Tbilisi
  - Cardioclinic Digomi Medical Center-, Tbilisi
  - David Metreveli Medical Centre Lt, Tbilisi
  - Emergency Cardiology Center by Academician G. Chapidze Ltd, Tbilisi
  - JSC Curatio, Tbilisi
  - LTD Adapti, Tbilisi
  - Ltd Georgian-Dutch Hospital, Tbilisi
  - LTD Israeli -Georgian Medical Research Clinic Healthycore, Tbilisi
  - Ltd Tbilisi Heart Center, Tbilisi
  - LTD Vitamed, Tbilisi
  - Mediclub Georgia, Tbilisi
  - Multiprofile Clinic Consilium Medulla LTD, Tbilisi
  - National Center for Diabetes Research, Tbilisi
  - Tbilisi Heart and Vascular Clinic Ltd, Tbilisi
  - The First Medical Center LTD, Tbilisi
  - VivaMedi, Tbilisi
- Germany (32):
  - Kardiologische Praxis Dr. med. univ. Wolfgang Jungmair, Bad Homburg
  - kfgn | Site Operations & Services GmbH - Berlin-Mitte, Berlin
  - Franziskus Hospital Berlin, Berlin
  - Diabetespraxis Dr. Braun, Berlin
  - Kardiologisch-Angiologische Praxis - Herzzentrum Bremen, Bremen
  - MVZ am Küchwald GmbH, Chemnitz
  - Gemeinschaftspraxis Diabeteszentrum Dortmund, Dortmund
  - St Johannes Hospital Dortmund, Dortmund
  - Kfgn | Site Operations & Services GmbH - Dresden, Dresden
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - ZKS - Zentrum Klinische Studien Sudbrandenburg GmbH, Elsterwerda
  - Katholisches Krankenhaus St. Johann Nepomuk, Erfurt
  - Klinisches Forschungszentrum Dr. Hagemann, Essen
  - Studienzentrum Bocholderstrasse, Essen
  - Zentrum für Klinische Studien (diabetes-falkensee.de), Falkensee
  - ClinPhenomics CVC GmbH, Frankfurt
  - Diabeteszentrum Hamburg West (DZHW) / Gemeinschaftspraxis Dr. Wendisch, Dr. Dahl und Prof. Dr. Aberle, Hamburg
  - St. Josefskrankenhaus Heidelberg GmbH, Heidelberg
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Velocity Clinical Research Leipzig GmBH, Leipzig
  - Diabetologikum DDG Ludwigshafe, Ludwigshafen
  - Kliniken Maria Hilf GmbH Krankenhaus St. Franziskus, Mönchengladbach
  - CDG Studienambulanz Dr. Hartard, München
  - Klinikum München Klinik Neuperlach, München
  - Praxis Drs. Haggenmiller/Jeserich, Nuremberg
  - RED-Institut GmbH, Oldenburg in Holstein
  - Praxis Reinfeld Mitte, Reinfeld
  - Herz Kreislauf Zentrum - Klinikum Hersfeld Rotenburg GmbH, Rotenburg (Wümme)
  - Studienzentrum Brinkum, Stuhr
  - Gemeinschaftspraxis Dr. med. Josef und Dr. med. Wilma Grosskopf, Wallerfing
  - Forschungszentrum Ruhr, Witten
  - INFO-MED Leipzig GmbH, Zwenkau
- Hungary (25):
  - Lausmed Kft, Baja
  - Tagore Medical Center, Balatonfüred
  - Dr Lakatos Ferenc Belgyogyaszati-Kardiologiai Maganrendelo, Békéscsaba
  - Qualiclinic Kft, Budapest
  - Semmelweis Egyetem - Szent Rokus Klinikai Tomb, Budapest
  - Del-pesti Centrumkorhaz, Budapest
  - MED-TIMA Kft, Budapest
  - Obudai Egeszsegugyi Centrum - Budapest, Budapest
  - Semmelweis Egyetem - Varosmajori Sziv es Ergyogyaszati Klinika, Budapest
  - Clinexpert Kft., Budapest
  - High Tech Medical Kft, Budapest
  - Belinus Bt, Debrecen
  - CRU Hungary Kft., Encs
  - Pharma4 Trial Kft, Gyöngyös
  - BKS Research Kft., Hatvan
  - Porcika Klinik, Hódmezővásárhely
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Pest M. Flór F. Kórház V. Belgy. Oszt, Kistarcsa
  - Kistarcsai Flor Ferenc Korhaz, Kistarcsa
  - IPR Hungary Kft, Miskolc
  - dr Vasas Szilard Haziorvosi Rendelo, Nyíregyháza
  - Medifarma-98 Kft, Nyíregyháza
  - dr Nagy Laszlo Kardiologiai Maganrendeles es Klinikai Vizsgalohely, Orosháza
  - Coromed SMO Kft, Pécs
  - Obudai Egeszsegugyi Centrum - Zalaegerszeg, Zalaegerszeg
- Israel (14):
  - Barzilai Medical Center, Ashkelon
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Hebrew University Medical Center - Cardiology - The Heart Institute, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galilee Medical Cente, Nahariya
  - Rabin Medical Center, Beilinson Hospital - Internal Medicine B, Petah Tikva
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - The BARUCH PADEH Medical Center, Poriya, Poria – Neve Oved
  - Kaplan Medical Center, Rehovot
  - Ziv Medical Center, Safed
  - Shamir Medical Center (Assaf Harofeh), Ẕerifin
- Italy (7):
  - Azienda Ospedaliero-Universitaria di Ferrara-Arcispedale Sant'Anna, Ferrara
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Santa Maria di Terni, Terni
- Japan (21):
  - Chiba University Hospital, Chiba
  - New Tokyo Heart Clinic, Chiba
  - Kokura Memorial Hospital, Fukuoka
  - Japan Community Health Care Organization Kyushu Hospital, Fukuoka
  - National Hospital Organization Takasaki General Medical Center, Gunma
  - Hiroshima Prefectural Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Hyogo Prefectural Harima-Himeji General Medical Center, Hyōgo
  - Ishikawa Prefectural Central Hospital, Ishikawa
  - Komatsu Municipal Hospital, Ishikawa
  - Public Central Hospital of Matto lshikawa, Ishikawa
  - Showa University Northern Yokohama Hospital, Kanagawa
  - Yokohama Minami Kyousai Hospital, Kanagawa
  - Niigata University Medical & Dental Hospital, Niigata
  - The Sakakibara Heart Institute of Okayama, Okayama
  - Sakurabashi Watanabe Hospital, Osaka
  - Saiseikai Senri Hospital, Osaka
  - National Cerebral and Cardiovascular Center Research Institute, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Osaka
  - Tokyo Saiseikai Central Hospital, Tokyo
  - Nihon University Itabashi Hospital, Tokyo
- Jordan (4):
  - Abdali Hospital, Amman
  - Istishari Hospital, Amman
  - Irbid Specialty Hospital, Irbid
  - Pharmaceutical Research Center -Jordan University of Science & Technology/King Abdulla University Hospital - Cardiology, Irbid
- Latvia (5):
  - Latgales Medical Center, Daugavpils
  - SIA ANIO, Daugavpils
  - D. Saulites-Kandevicas Private Practice, Liepāja
  - Pauls Stradins Clinical University Hospital Riga, Riga
  - Vidzemes Hospital, Valmiera
- Netherlands (21):
  - Academic Medical Center - Department of Vascular Medicine, Amsterdam
  - Ziekenhuis Rijnstate, Arnhem
  - Rode Kruis Ziekenhuis, Beverwijk
  - Reinier de Graaf Gasthuis, Delft
  - Het Van Weel-Bethesda Ziekenhuis, Dirksland
  - Albert Schweitzer Ziekenhuis - Location Dordrecht, Dordrecht
  - Ziekenhuis Gelderse Vallei, Ede
  - Maxima Medisch Centrum, Eindhoven
  - Groene Hart Ziekenhuis, Gouda
  - St. Jansdal Ziekenhuis, Harderwijk
  - Elkerliek Ziekenhuis - Locatie Helmond, Helmond
  - Treant Zorggroep, Hoogeveen
  - Leids Universitair Medisch Centrum, Leiden
  - Stichting Radboud Universitair Medisch Centrum, Nijmegen
  - Canisius-Wilhelmina Ziekenhuis (CWZ), Nijmegen
  - Franciscus Gasthuis & Vlietland - Locatie Gasthuis, Rotterdam
  - HMC Westeinde, The Hague
  - Diakonessenhuis - Locatie Utrecht, Utrecht
  - VieCuri Medisch Centrum, Venlo
  - Zaans Medisch Centrum, Zaandam
  - Albert Schweitzer Ziekenhuis - Location Zwijndrecht, Zwijndrecht
- Poland (48):
  - CENTRUM MEDYCZNE INTERCOR Sp. z o.o., Bydgoszcz
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz
  - Centrum Medyczne Kermed - Renata Bijata-Bronisz I Ewa Kowalinska Spólka Jawna, Bydgoszcz
  - DIAB Serwis Popenda Spólka Jawna, Chorzów
  - NZOZ Twoje Zdrowie EL Sp. z o.o., Elblag
  - Indywidualna Specjalistyczna Praktyka Lekarska dr n. med. Adam Grzybowski, Gdansk
  - Uniwersyteckie Centrum Kliniczne, I Klinika Kardiologii, Gdansk
  - Indywidualna Specjalistyczna Praktyka Lekarska w Dziedzinie Kardiologii, lek. med. Krzysztof Cymerman, Gdynia
  - Samodzielny Publiczny Specjalistyczny Szpital Zachodni im. Jana Pawla II, Grodzisk Mazowiecki
  - Centrum Medyczne Pratia Katowice, Katowice
  - SALVIA Lekston i Madej s.j., Katowice
  - Silmedic Sp. z o.o., Katowice
  - Ewa Mirek-Bryniarska Specjalistyczna Praktyka Lekarska, Krakow
  - Pratia MCM Krakow, Krakow
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II - Oddzial Kliniczny Kardiologii Interwencyjnej z Pododdzialem Intenyswengo Nadzoru Kardiologicznego, Krakow
  - Centrum Medyczne ZDROWA, Krakow
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - ETG Lodz - Santa Sp. z. o.o., Lodz
  - FutureMeds Lodz, Lodz
  - INSTYTUT CENTRUM ZDROWIA MATKI POLKI - Klinika Kardiologii i Wad Wrodzonych Doroslych, Lodz
  - Indywidualna Specjalistyczna Praktyka Lekarska Wlodzimierz Kus, Lodz
  - Clinical Best Solutions - Lublin, Lublin
  - KO - MED Centra Kliniczne Lublin II, Lublin
  - ETG Lublin - Pro Life Medica Sp. z o.o, Lublin
  - Szpital Sw. Anny w Miechowie, Miechów
  - Pomorskie Centra Kardiologiczne Sp. z o.o., SKA - Mragowo, Mrągowo
  - Futuremeds Olsztyn, Olsztyn
  - Ostrowieckie Centrum Medyczne spólka cywilna Anna Olech-Cudzik, Ostrowiec Świętokrzyski
  - ZOZ w Olawie, Oddzial Chorob Wewnetrznych, Oława
  - Centrum Medyczne OMEDICA Jaroslaw Opiela i Beata Opiela s. j., Poznan
  - NZOZ Neuro-Kard - Ilkowski i Partnerzy Spólka Partnerska Lekarzy, Poznan
  - Aka-Med Centrum Spólka Z Ograniczona Odpowiedzialnoscia, Ruda Śląska
  - ETG Siedlce- Lukmed 2 Sp. z o.o., Siedlce
  - ETG Skierniewice - ClinMedica Research Sp. z o.o., Skierniewice
  - NZOZ Pro Cordis Sopockie Centrum Badan Kardiologicznych, Sopot
  - Nowe Zdrowie-Ck Kieltucki i Wspolnicy Spolka Jawna, Staszów
  - Osrodek Badan Klinicznych LabMed Agnieszka Karczmarczyk, Filip Karczmarczyk Spólka Cywilna, Szczecin
  - Prywatny Gabinet Lekarski Jacek Gessek, Torun
  - FutureMeds Warszawa Centrum, Warsaw
  - ETG Warszawa- MCM Polimedica 2 Sp. z o.o., Warsaw
  - FutureMeds Targowek, Warsaw
  - Clinical Best Solutions Sp. z.o.o Spolka Komandytowa, Warsaw
  - Narodowy Instytut Kardiologii Stefana kardynala Wyszynskiego - Panstwowy Instytut Badawczy, Poradnia Prewencji i Leczenia Chorob Metabolicznych, Zaklad Epidemiologii, Prewencji Chorób Ukladu Krazeni, Warsaw
  - FutureMeds Sp. z o.o, Wroclaw
  - 4 Wojskowy Szpital Kliniczny z Poliklinika Samodzielny Publiczny ZOZ we Wroclawiu, Wroclaw
  - Wroclawska Grupa Medyczna Pankiewicz Spolka Jawna, Wroclaw
  - ETG Zamosc - Pro Life Medica Sp. z o.o, Zamość
  - KO - MED Centra Kliniczne Sp. z o.o., Osrodek Badan Klinicznych w Zamosciu, Zamość
- Slovakia (24):
  - Stredoslovensky ustav srdcovych a cievnych chorob, a.s., Banská Bystrica
  - Alian, s.r.o., Kardiologicka ambulancia, Bardejov
  - DIADA s.r.o., Bardejov
  - Thyreomedical s.r.o., Bardejov
  - Medispektrum s.r.o., Diabetologicka a metabolicka ambulancia, Bratislava
  - Univerzitna nemocnica Bratislava, Bratislava
  - Kardiologicka ambulancia NsP, n.o., Brezno
  - JM-INTERNA, s.r.o., Ambulancia vnutorneho lekarstva, Dolný Kubín
  - Cardio D&R, S.R.O. Kosice, Košice
  - Human-Care s.r.o, Košice
  - Medical group Kosice, s.r.o. - Kardiologicka a Interna ambulancia, Košice
  - KardioLEV s. r. o., Levoča
  - Kardiomed s.r.o., Lučenec
  - KARDIO 1 s.r.o., Lučenec
  - Interna a diabetologicka ambulancia - IN - DIA s.r.o., MUDr. Livia Tomasova, Lučenec
  - Univerzitna nemocnica Martin, Martin
  - Medi M and M sro, Moldava nad Bodvou
  - Kardiocentrum Nitra s.r.o., Nitra
  - Medical KG, s.r.o. - Ambulancia vnutorneho lekarstva, Piešťany
  - Medispol, s.r.o., Prešov
  - Tatratrial s.r.o, Rožňava
  - Interna SK, s.r.o., Kardiologicka a interna ambulancia, Svidník
  - JAL s.r.o., Trnava
  - Medivasa, s.r.o., Angiologicka a kardiologicka ambulancia, Žilina
- South Africa (7):
  - Iatros International, Bloemfontein
  - Tiervlei Trial Centre (TTC), Cape Town
  - TREAD Research - Department of Cardiology, Cape Town
  - WCR - Bara Cardiology, Johannesburg
  - Dr JM Engelbrecht Trial Site, Somerset West
  - Helderberg Research Institute, Somerset West
  - Mediclinic Victoria, Tongaat
- Spain (16):
  - Hospital Universitario de A Coruna, A Coruña
  - Hospital General Universitario de Alicante Dr. Balmis, Alicante
  - Hospital Universitario Torrecardenas, Almería
  - Hospital del Mar, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Joan XXIII de Tarragona, Tarragona
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Alvaro Cunqueiro, Vigo
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (27):
  - Atlantic Medical Group, Penzance, Cornwall
  - Mounts Bay Medical, Penzance, Cornwall
  - Ulster Hospital, Belfast
  - FutureMeds - Soho Road Health Centre, Birmingham
  - Birmingham Heartlands Hospital, Birmingham
  - Waterloo Medical Centre, Blackpool
  - University Hospital of Wales, Cardiff
  - FutureMeds - Ely Bridge Surgery, Cardiff
  - Darlington Memorial Hospital, Durham
  - Panthera - London North, Enfield
  - Fowey River Practice, Fowey
  - Panthera - Glasgow, Glasgow
  - Futuremeds - CPS Research, Glasgow
  - Hounslow Medical Centre, Hounslow
  - St. Bartholomew's Hospital, London
  - The Good Practice, London
  - Chelsea and Westminster Hospital, London
  - Luton and Dunstable University Hospital, Luton
  - FutureMeds - Bridle Road Clinic, Metropolitan Borough of Wirral
  - Beacon Medical Group, Plymouth
  - Craigavon Area Hospital, Portadown
  - Panthera - Preston, Preston
  - Panthera - Manchester, Rochdale
  - Queens Hospital, Romford
  - Panthera - Sheffield, Sheffield
  - Sandwell General Hospital, West Bromwich
  - Worcestershire Royal Hospital, Worcester

IPD SHARING:
Plan to Share IPD: No